CLINICAL TRIAL: NCT07194707
Title: The Effect of Operating Room Environmental Noise on BIS and Hemodynamics in Patients Under General Anesthesia: A Prospective Observational Study
Brief Title: Effect of Operating Room Noise on BIS and Hemodynamics Under General Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine OZCAN, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: SOUNDM3419
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: General Anesthesia; Hemodynamics; Noise Exposure
Keywords: Anesthesia, General; Operating Rooms; Monitoring, Intraoperative; Hemodynamics; Bispectral Index (BIS); Noise Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 (Noisy Group): Patients exposed to average OR noise level >65 dB during general anesthesia.
  Interventions: Other: Intraoperative Noise Monitoring
- 2 (Quiet Group): Patients exposed to average OR noise level <55 dB during general anesthesia.
  Interventions: Other: Intraoperative Noise Monitoring

INTERVENTIONS:
Other: Intraoperative Noise Monitoring — Noise levels will be passively measured during surgery using a calibrated sound level meter (CEM DT-8850) placed near the patient's head. Measurements will be taken every 10 minutes without physical contact or interference with clinical care. The procedure is purely observational and does not modify anesthesia or surgical practice.
  Other Names: CEM DT-8850 Sound Level Meter; Operating Room Noise Measurement

SUMMARY:
This prospective observational study aims to evaluate the impact of operating room noise on bispectral index (BIS) and hemodynamic parameters in patients undergoing general anesthesia. Environmental noise in operating rooms, often overlooked, may influence anesthesia depth, patient safety, and physiological stability. A total of 70 adult patients (ASA I-II, 18-65 years, elective surgery under general anesthesia) will be enrolled at Başakşehir Çam and Sakura City Hospital. Patients will be categorized into two groups based on intraoperative average noise levels: noisy group (>65 dB) and quiet group (<55 dB). Noise levels will be measured every 10 minutes using a CEM DT-8850 sound level meter, BIS will be recorded every 10 minutes, and hemodynamic variables (systolic, diastolic, mean arterial pressure, and heart rate) will be recorded every 5 minutes.

Primary outcome is the correlation between mean intraoperative noise levels (LAeq) and BIS values during the maintenance phase of anesthesia. Secondary outcomes include the relationship between noise characteristics (e.g., device-related, human-related, alarms, media) and hemodynamic stability, as well as surgical branch-related noise classifications (high, moderate, low). The study is non-interventional, with no additional risk to participants beyond standard clinical monitoring. Findings are expected to provide evidence on the role of environmental noise in anesthesia quality, inform operating room organization, and contribute to patient safety improvements.

DETAILED DESCRIPTION:
Operating room (OR) noise is a common but underestimated environmental factor that may affect both patients and medical staff. In patients under general anesthesia, excessive noise may influence depth of anesthesia, physiological stability, and recovery outcomes.This prospective observational study will investigate the correlation between intraoperative noise levels and bispectral index (BIS) values, as well as hemodynamic parameters (systolic, diastolic, and mean arterial pressure, and heart rate). Seventy adult patients undergoing elective surgery under general anesthesia will be monitored. Noise levels will be measured every 10 minutes with a calibrated sound level meter (CEM DT-8850), while BIS and hemodynamic parameters will be recorded at 10-minute and 5-minute intervals, respectively. Additionally, the type of noise (device-related, human-related, alarms, media) and the surgical branch (classified into high, moderate, or low noise categories) will be documented. Data will be analyzed to determine whether environmental noise correlates with BIS fluctuations and hemodynamic stability. The study is observational only and involves no intervention beyond standard anesthesia practice. Results are expected to raise awareness of environmental influences on anesthesia management and provide recommendations for OR organization to enhance patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70
* ASA (American Society of Anesthesiologists) physical status score I-II
* Scheduled for elective surgery
* To be undergoing general anesthesia
* Having signed the informed consent form to participate in the study

Exclusion Criteria:

* Hearing impairment or ear pathology
* History of neurological disease (epilepsy, stroke, dementia, etc.)
* Use of psychiatric medications (anxiolytics, antidepressants, antipsychotics, etc.)
* Indications for emergency surgery
* Planned spinal or epidural anesthesia
* Conditions unsuitable for BIS monitoring
* Cognitive impairment preventing informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-70 years undergoing elective surgery under general anesthesia at Başakşehir Çam and Sakura City Hospital will be included. Eligible participants must have ASA physical status I-II, be cognitively able to provide informed consent, and scheduled for surgeries lasting up to 2 hours. Both male and female patients will be enrolled without restriction. Only elective (non-emergency) procedures are considered. Surgeries from multiple specialties (orthopedics, neurosurgery, cardiovascular, general surgery, gynecology, urology, ophthalmology, otolaryngology, plastic surgery, dermatology) will be included, representing high, moderate, and low noise exposure categories.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between intraoperative noise levels and BIS values | 10-minute intervals intraoperative period
  Relationship between mean intraoperative noise levels (LAeq, dB(A)) and mean Bispectral Index (BIS) values during the maintenance phase of general anesthesia.

SECONDARY OUTCOMES:
Relationship between intraoperative noise levels and hemodynamic parameters | Intraoperative period
  Association between average intraoperative noise level (LAeq, dB(A)) and hemodynamic variables (systolic blood pressure, diastolic blood pressure, mean arterial pressure, and heart rate). Hemodynamic parameters will be recorded at 5-minute intervals, while noise levels will be measured at 10-minute intervals.
Effect of noise source type on BIS and hemodynamic stability | Intraoperative period.
  Evaluation of whether noise source categories (device-related, human-related, alarms, media) are associated with changes in BIS and hemodynamic parameters. Noise type will be recorded by independent observer every 10 minutes.
Comparison of BIS and hemodynamic outcomes across surgical branches | Intraoperative period.
  Surgical specialties will be classified into high, moderate, or low noise categories. BIS and hemodynamic data will be compared across these groups.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Ozcan, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and confidentiality concerns. Only aggregated results will be published in scientific journals and conferences.

REFERENCES:
- [Background] Li X, Li J, Xu Z, Shang Y, Shi H. Effects of Operating Room Noise on Patient Outcomes and Medical Staff: A Systematic Review. Noise Health. 2025 May-Jun 01;27(126):246-254. doi: 10.4103/nah.nah_175_24. Epub 2025 Jun 26. PMID 40574295
- [Background] You S, Xu F, Zhu X, Qin S, Zheng X, Tao C, Wu Y, Chen Y, Shu B, Huang H, Duan G. Effect of intraoperative noise on postoperative pain in surgery patients under general anesthesia: evidence from a prospective study and mouse model. Int J Surg. 2023 Dec 1;109(12):3872-3882. doi: 10.1097/JS9.0000000000000672. PMID 37598384
- [Background] Jeyaraman M, Jeyaraman N, Yadav S, Nallakumarasamy A, Iyengar KP, Jain V. Impact of Excessive Noise Generation in Orthopaedic Operating Theatres: A Comprehensive Review. Cureus. 2024 Feb 19;16(2):e54469. doi: 10.7759/cureus.54469. eCollection 2024 Feb. PMID 38510860
- [Background] Louis M, Grabill N, Strom P, Gibson B. Leading Through Noise: Operating Room Noise Challenges for Staff and Leadership Techniques to Ensure Optimal Operational Performance. Cureus. 2024 Sep 17;16(9):e69569. doi: 10.7759/cureus.69569. eCollection 2024 Sep. PMID 39421089